CLINICAL TRIAL: NCT05076838
Title: An Open-Label, Single-Dose, Pharmacokinetics Study of VALTOCO® With Open-Label Safety Period in Pediatric Subjects With Epilepsy
Brief Title: Pharmacokinetics Study of VALTOCO® in Pediatric Subjects With Epilepsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurelis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAZ.001.08
Record Dates: First submitted 2021-09-15; First posted 2021-10-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valtoco In Pediatric Subjects with Epilepsy (Experimental): 5 mg, 10 mg, or 15 mg dose of intranasal VALTOCO will be administered based on the subject's body weight.
  Interventions: Drug: Diazepam Nasal Spray [Valtoco]

INTERVENTIONS:
Drug: Diazepam Nasal Spray [Valtoco] — 5 mg, 10 mg, or 15 mg dose of intranasal VALTOCO will be administered based on the subject's body weight.

SUMMARY:
This is a Phase 1/2a, open-label, single-dose, PK study of VALTOCO with open-label safety period in pediatric epilepsy subjects age 2 to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of epilepsy and, in the opinion of the Investigator, may need benzodiazepine intervention for seizure control.
* Subjects having either partial or generalized epilepsy with motor seizures or seizures with clear alteration of awareness, for which rescue medications have been used at least once in the last 3 months or in the opinion of the investigator, may need a benzodiazepine intervention for seizure control 1-2 times every 3 months on average.

Exclusion Criteria:

* Subjects whose body weight are < 6 kg or > 33 kg.
* Subject is undergoing intracranial electroencephalogram (EEG) monitoring.
* In the opinion of the investigator, a history of clinically significant medical history that would jeopardize the safety of the subject or impact the validity of the study results (such as significant gastrointestinal, renal, nasal polyps or any nasal passage abnormality that could interfere with nasal spray administration.
* Subject has had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.
* Inadequate or difficult venous access that may jeopardize the quality or timing of the PK samples.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of diazepam after intranasal VALTOCO administered to subjects with epilepsy 2 to 5 years of age | 0-6 hours

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Northwest Florida Clinical Research Group, LLC., Gulf Breeze, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Research Institute, Orlando, Florida
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Missouri Women & Children's Hospital, Columbia, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Boston Children's Health Physicians, Hawthorne, New York
  - University of Rochester, Rochester, New York
  - Duke University Hospital, Durham, North Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia